CLINICAL TRIAL: NCT02711605
Title: Clinical Evaluation of the UltraShape Device for Non-Invasive Fat Reduction in the Male Breast (Pseudogynecomastia)
Brief Title: UltraShape Device for Non-Invasive Fat Reduction in the Male Breast (Pseudogynecomastia)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never got underway due to sponsor re-organization.
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DHF21271
Record Dates: First submitted 2016-03-13; First posted 2016-03-17 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Gynecomastia; Male Breast Enlargement
Keywords: ultrasound; fat
MeSH Terms: conditions — Gynecomastia; Platelet Glycoprotein IV Deficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Unilateral UltraShape treatment (Experimental): One side of the chest (left or right breast) will be treated with the UltraShape focused ultrasound device, while the opposite will serve as an untreated control.
  Interventions: Device: UltraShape focused ultrasound device
- Bilateral UltraShape treatment (Experimental): Both sides of the chest (right and left breasts) will be treated with the UltraShape focused ultrasound device.
  Interventions: Device: UltraShape focused ultrasound device

INTERVENTIONS:
Device: UltraShape focused ultrasound device — 3 biweekly focused ultrasound treatments to the male chest with UltraShape.
  Other Names: Contour I

SUMMARY:
Male volunteers who suffer from Pseudogynecomastia and seek noninvasive breast fat reduction will be enrolled into two arms to receive three biweekly UltraShape treatments.

DETAILED DESCRIPTION:
Up to 40 adult male volunteers, who suffer from Pseudogynecomastia, and seek noninvasive breast fat reduction will be enrolled at up to three investigational sites. Eligible subject will be divided into one of the two treatment arms: Arm 1: Subjects will be treated on one side of the breast, while the opposite side will serve as control - Up to 20 subjects; Arm 2: Subjects will be treated on both sides of the breast - Up to 20 subjects. Subjects will receive 3 bi-weekly treatments (at 2-week intervals) with the UltraShape device.

Subjects will return for 3 follow-up visits post last treatment (Tx.3): four weeks follow-up (4wk FU), eight weeks follow-up (8wk FU) and 12 weeks follow-up (12wk FU) for total expected study duration of 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent to participate in the study
2. Male subjects, 18 -70 years of age at the time of enrollment
3. BMI interval: BMI ≥ 22 and ≤30 (normal to overweight, but not obese)
4. Fat thickness of at least 1.5 cm in the treated area (breast) as measured by calibrated caliper.
5. Subject has clearly visible, palpable, excess fatty tissue in their breast area, and minimal fibrous tissue.
6. Subject agrees to maintain their weight (i.e., within 3% weight change) by not making any major changes in their diet or lifestyle during the course of the study.
7. General good health confirmed by medical history and skin examination of the treated area.
8. Willing to follow the treatment and follow-up schedule and post-treatment care instructions.
9. Willing to have photographs and images taken of the treated areas to be used, de-identified in evaluations, publications and presentations.

Exclusion Criteria:

1. History of hypertension, ischemic heart disease, valvular heart disease, congestive heart failure, pacemaker/defibrillator.
2. Known hyperlipidemia, diabetes mellitus, hepatitis, liver disease, HIV positive status, blood coagulopathy or excessive bleeding, autoimmune or connective tissue disease.
3. Having or undergoing any form of treatment for active cancer, or having a history of skin cancer or any other cancer in the areas to be treated, including presence of malignant or pre-malignant pigmented lesions.
4. Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator.
5. Having a permanent implant in the treated area, such as metal plates or an injected chemical substance such as silicone.
6. Having undergone any other surgery in the treated areas within 12 months of treatment or during the study, including liposuction.
7. Previous body contouring procedures in the treatment area within 12 months.
8. History of skin disease in the treatment area, known tendency to form keloids or poor wound healing.
9. Suffering from significant skin conditions in the treated areas or inflammatory skin conditions, including, but not limited to, open lacerations or abrasions and active cold sores or herpes sores prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course.
10. Skin lesions in the treatment area other than simple nevi on physical examination (e.g., atypical nevus, tattoo, abrasions) including depressed scars in the treatment area.
11. Very poor skin quality (i.e., severe laxity) according to the investigator decision.
12. Obesity (BMI >30).
13. Unstable weight within the last 6 months (i.e., 3% weight change in the prior six months).
14. Inability to comply with circumference measurement procedure (e.g., inability to hold breath for the required duration).
15. Fat thickness lower than 2.5 cm after strapping at the treated area.
16. Participation in another clinical study involving same anatomical areas within the last 6 months (or 30 days in case different anatomical areas were treated in previous trial/s).
17. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.
18. Personal history of previous breast malignancy.
19. Subject is taking any medication which could cause abnormal breast enlargement - including but not limited to: digoxin, furosemide, gonadotropins, clomiphene, phenytoin, and exogenous testosterone, ketoconazole, metronidazole, alkylating agents, cisplatin, spironolactone, cimetidine, flutamide, finasteride, etomidate, isonicotinic acid hydrazide, methyldopa, busulfan, tricyclic antidepressants, diazepam, penicillamine, omeprazole, phenothiazines, calcium channel blockers, angiotensin-converting enzyme (ACE) inhibitors.
20. Subject has history of the following medical conditions: Klinefelter syndrome, Congenital anorchia, Testicular trauma, Testicular torsion, Viral orchitis, Kallmann syndrome , Pituitary tumors, Malignancies that increase the serum level of hCG (eg, large cell lung cancer, gastric carcinoma, renal cell carcinoma, hepatoma), Renal failure, Hyperthyroidism, Malnutrition, Androgen insensitivity syndrome, Five-alpha-reductase deficiency syndrome.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03-13 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2017-12-06 (Actual)

PRIMARY OUTCOMES:
Reduction in breast fat thickness after 3 treatments compared to baseline | 12 weeks after 3rd treatment (16 weeks)
  Average reduction in breast fat thickness after 3 treatments compared to baseline, as measured by ultrasound imaging

SECONDARY OUTCOMES:
Reduction in breast fat thickness on treated side compared to control side | 12 weeks after 3rd treatment (16 weeks)
  Average reduction in breast fat thickness on treated side compared to control side, as measured by ultrasound imaging (Arm 1 only)
Reduction in breast/chest circumference after 3 treatments compared to baseline | At 4-week, 8-week and 12-week follow-ups
  Average reduction in breast/chest circumference after 3 treatments compared to baseline, as measured by measuring tape (Arm 2 only)
Reduction in breast fat thickness compared to baseline | At 4-week, 8-week and 12-week follow-ups
  Average reduction in breast fat thickness compared to baseline, as measured by skin caliper
Reduction in breast fat thickness on treated side compared to control side | At 4-week, 8-week and 12-week follow-ups
  Average reduction in breast fat thickness on treated side compared to control side, as measured by skin caliper (Arm 1 only)

OTHER OUTCOMES:
Number of participants with adverse events | through study duration up to 1 year
  The number of adverse events, severity, intervention and outcome, as reported on adverse event forms

CONTACTS AND LOCATIONS:
Overall Officials: Shlomit Mann, MA, Study Director — Syneron Medical

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Moreno-Moraga J, Valero-Altes T, Riquelme AM, Isarria-Marcosy MI, de la Torre JR. Body contouring by non-invasive transdermal focused ultrasound. Lasers Surg Med. 2007 Apr;39(4):315-23. doi: 10.1002/lsm.20478. PMID 17457840